CLINICAL TRIAL: NCT04476771
Title: Cultivating Well-being Beyond Symptomatology in Subclinical Paranoia: A Randomized Controlled Trial
Brief Title: Cultivating Well-being in Subclinical Paranoia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Carmen Valiente Ots, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ComplutenseMadrid
Record Dates: First submitted 2017-10-10; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Wellbeing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + waiting list (No Intervention): Feliz-Mente (third generation psychotherapy):The intervention is delivered in a group format with a total of 12 sessions and a maximum of 10 patients per group. The protocol consists of specific exercises: 1: welcome and identification of emotions, 2: identification and amplification of positive emotions, 3: regulation of negative emotions, 4: gratitude, 5: forgiveness, 6: self-compassion, 7: personal strengths, 8: loving-kindness and positive interpersonal relationships, 9: values, 10: purpose of life, 11: resilience, 12: keeping the change and farewell party.
- TAU + Feliz-Mente Intervention (Experimental): Feliz-Mente (third generation psychotherapy):The intervention is delivered in a group format with a total of 12 sessions and a maximum of 10 patients per group. The protocol consists of specific exercises: 1: welcome and identification of emotions, 2: identification and amplification of positive emotions, 3: regulation of negative emotions, 4: gratitude, 5: forgiveness, 6: self-compassion, 7: personal strengths, 8: loving-kindness and positive interpersonal relationships, 9: values, 10: purpose of life, 11: resilience, 12: keeping the change and farewell party.
  Interventions: Behavioral: Feliz-Mente (third generation psychotherapy)

INTERVENTIONS:
Behavioral: Feliz-Mente (third generation psychotherapy) — The intervention is delivered in a group format with a total of 12 sessions and a maximum of 10 patients per group. The protocol consists of specific exercises: 1: welcome and identification of emotions, 2: identification and amplification of positive emotions, 3: regulation of negative emotions, 4: gratitude, 5: forgiveness, 6: self-compassion, 7: personal strengths, 8: loving-kindness and positive interpersonal relationships, 9: values, 10: purpose of life, 11: resilience, 12: keeping the change and farewell party.
  Arms: TAU + Feliz-Mente Intervention

SUMMARY:
The intervention is called Feliz-Mente, with third generation therapy components that aims to improve wellbeing and self-enhancement. Without intervening directly on the symptoms, it is expected to increase positive experiences, the use of personal strengths and positive relationships, and aims to build a more meaningful self-narrative in persons with subclinical paranoia. Feliz-Mente is a group intervention of 12 sessions in which participants are expected to perform exercises during and between sessions by the use of a mobile application to improve treatment adherence and daily practice. The design for the present study is a randomized controlled trial, which compares the post-intervention measures of the experimental group (group receiving the intervention and the daily use of a mobile application of the program) with the post-intervention measures of the control group (treatment as usual + waiting list).

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 35 years old
* At least two standard deviations above mean on the scales of distress, suspicion and /or interpersonal sensitivity in the SCL-90 questionnaire.

Exclusion Criteria:

* Participants with borderline personality disorder
* Participants with substance use disorders and /or
* Participants with severe cognitive impairment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Change from Well-being at 12 weeks, 3 months and 12 months | Change baseline, 12 weeks, 3 months and 12 months
  Psychological Well-Being Scales (Ryff, 1995)
Change from Well-being at 12 weeks, 3 months and 12 months | Change baseline, 12 weeks, 3 months and 12 months
  Satisfaction with life Scale ( Diener et al. 1985)

SECONDARY OUTCOMES:
Change from Well-beingDistress at 12 weeks, 3 months and 12 months | Change baseline, 12 weeks, 3 months and 12 months
  Hospital Anxiety and Depression Scale (Bjelland et al. 2002)
Change from self-esteem at 12 weeks, 3 months and 12 months | Change baseline, 12 weeks, 3 months and 12 months
  Implicit self-esteem version: Go/No-Go Association Task (Nosek & Banaji, 2001)
Change from self-esteem at 12 weeks, 3 months and 12 months | Change baseline, 12 weeks, 3 months and 12 months
  Rosenberg self-esteem scale (Rosenberg, 1965)
Change from Attachment at 12 weeks, 3 months and 12 months | Change baseline, 12 weeks, 3 months and 12 months
  Relationship Questionnaire (Bartholomew and Horowitz, 1991)
Change from Paranoid ideation at 12 weeks, 3 months and 12 months | Change baseline, 12 weeks, 3 months and 12 months
  Persecutory Ideation Questionnaire(McKay, Langdon and Coltheart, 2006)
additional Outcome Measures Experience of trauma events | baseline
  Life Events Checklist for DSM-5 (Gray, 2004)

CONTACTS AND LOCATIONS:
Locations (1):
- Carmen Valiente, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code